CLINICAL TRIAL: NCT02748369
Title: In Vivo Assessment of the Tricarboxylic Acid Cycle Flux in the Muscle and Splanchnic Bed of Humans: A Pilot Study
Brief Title: In Vivo Assessment of Cellular Metabolism in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: K. Sreekumaran Nair (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, K. Sreekumaran Nair, M.D., P.h.D. ; Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-000085; U24DK100469 (NIH)
Record Dates: First submitted 2016-04-12; First posted 2016-04-22 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Normal Cellular Metabolism
Keywords: TCA cycle flux; in vivo measurements; Stable isotopes; Arteriovenous balance; Metabolome; Proteome; Exosomes
MeSH Terms: interventions — Somatostatin; Somatostatin-28; Glucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No somatostatin and glucagon infusions
- Intervention Group (Active Comparator): Somatostatin and glucagon infusions
  Interventions: Drug: Somatostatin; Drug: Glucagon

INTERVENTIONS:
Drug: Somatostatin — Somatostatin infusion to create a low insulin state.
  Other Names: growth hormone-inhibiting hormone
  Arms: Intervention Group
Drug: Glucagon — Glucagon infusion in the setting of ongoing somatostatin.
  Other Names: Glucagen
  Arms: Intervention Group

SUMMARY:
This is a pilot study to establish an arterial venous methodology to measure the activity of the TCA cycle or flux directly in tissues of human beings. It will also perform correlative studies to study the proteome, metabolome, oxygen consumption, carbon dioxide production and exosomes derived from the arterial venous supply of tissues with correlation to the TCA cycle activity.

DETAILED DESCRIPTION:
The tricarboxylic (TCA) or Krebs cycle is the "central hub of cellular metabolism" that takes place within the mitochondria. It is a series of sequential chemical reactions that generate cellular energy in the form of ATP. In addition, the cycle provides intermediate metabolites that are utilized in the biosynthesis of amino acids and fatty acids as well as reducing agents such as nicotinamide adenine dinucleotide (NADH) and flavin adenine dinucleotide (FADH2) that are used in numerous biochemical reactions. The dysfunction of the TCA cycle is recognized for its association in neurodegenerative and cardiovascular diseases, metabolic syndromes, tumorigenesis and aging. Hence, being able to measure the activity or flux of the TCA cycle either in vitro or in vivo holds significant clinical significance. Almost all studies are based on in vitro approaches except NMRS based studies that involve multiple non-validated assumptions.

Various stable isotope labeling studies have been used to estimate the TCA cycle flux by measuring one or more labelled intermediate metabolites within the cycle. Unfortunately, these labelled intermediates are often present through only partial segments of the cycle due to exchange, anaplerosis (entrance into the cycle), cataplerosis (export out of the cycle) or incomplete cycling. Though these previous isotope labeling studies of the TCA cycle flux were qualitatively informative, many were quantitatively inaccurate due to unexpected dilutions of the TCA cycle intermediates arising from unlabeled precursors.

This is a pilot study to establish a novel methodology using mass-isotopomer flux analysis after infusions of 2-13C-Acetate, 2-15N-Glutamine and D5-phenylalanine to measure the in vivo TCA cycle flux in tissues of human beings. This study will simultaneously determine the validity of measuring the TCA cycle flux in tissue indirectly through dynamic differences in enrichment of labelled TCA cycle intermediates between arterial and venous blood supplies of that particular tissue bed (i.e. arteriovenous model or A-V balance technique). We propose to measure the rates of the different metabolic reactions within the TCA cycle by tracing the position-specific 13C and 15N transfer between the intermediate metabolites in order to characterize the oxidative, anaplerotic, cataplerotic and exchange rates across the TCA cycle. The use of 2-15N-Glutamine will specifically allow us to determine the rate of glutamine entry into the cycle via its conversion to glutamate, thus providing a more accurate quantification of the TCA flux.

This methodology will be validated in the setting of controlled physiologic perturbations in human study participants such as low endogenous insulin levels alone or in combination with high glucagon levels.

Finally, correlative studies evaluating the mitochondrial activity in the skeletal muscle tissue, the oxygen consumption in the skeletal and splanchnic tissue beds, the role of circulating exosomes derived from the arteriovenous circulation of the skeletal and splanchnic tissue beds and the changes in the whole body metabolome will also be performed:

* First, mitochondrial respiration will be measured by high resolution respirometry (Oxygraph, Oroboros Instruments, Innsbruck, Austria) using a stepwise protocol to evaluate various components of the electron transport system. Protein content of the mitochondrial suspension will be measured using a colorimetric assay (Pierce 660-nm Protein Assay). Oxygen flux rates will be expressed per tissue-wet weight and per milligram of mitochondrial protein.
* Secondly, reactive oxygen species (ROS) emissions will also be evaluated on all skeletal muscle tissue samples. Briefly, a Fluorolog 3 (Horiba Jobin Yvon) spectrofluorometer with temperature control and continuous stirring will be used to monitor Amplex Red (Invitrogen) oxidation in freshly isolated mitochondrial suspensions obtained from the skeletal muscle biopsies. Amplex Red oxidation will be measured in the presence of glutamate (10 mmol/L), malate (2 mmol/L), and succinate (10 mmol/L). The fluorescent signal will be corrected for background auto-oxidation and calibrated to a standard curve. The H2O2 production rates will be expressed relative to mitochondrial protein.
* Third, simultaneous assessments of the oxygen consumption and carbon dioxide production will be determined through blood gas measurements from the arteriovenous samples obtained from the splanchnic and skeletal muscle tissue beds. These assessments will be performed at all three time points of blood sample assessments and correlated with the measured TCA cycle flux in their respective tissue beds.
* Circulating exosomes will also be derived from the arteriovenous samples of the splanchnic and skeletal muscle tissue beds to determine its intra-exosome proteome and metabolome and its relationship with the TCA cycle flux in their respective tissue beds. Incorporation of D5-phenylalanine will help trace the protein formation in the exosomes.
* Finally, changes in the whole body metabolome and proteome determined via the arteriovenous samples obtained from the splanchnic and skeletal muscle tissue beds will also be performed and correlated with the TCA cycle flux in their respective tissue beds.

ELIGIBILITY:
INCLUSION CRITERIA:

* Ages 18-45
* Able to provide written consent

EXCLUSION CRITERIA:

* Diabetes mellitus or impaired fasting glucose levels (fasting blood glucose >110mg/dl).
* Renal Failure
* Pregnancy
* Steroid use
* Muscle Disease
* Liver Disease
* Major Depression
* Anemia
* H/O alcohol use
* Medications other than OCPs
* BMI of 30 or greater

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
In Vivo TCA cycle flux in skeletal muscle and splanchnic tissue | 12 hours
  Normal healthy study participants will receive an initial priming dose followed by a continuous infusion of 2-13C-Acetate, 2-15N-Glutamine and D5-Phenylalanine in order to achieve steady state enrichment of 13C and 15N in their system. Serial arteriovenous blood samples will be obtained from the femoral artery, femoral vein and hepatic vein and serial skeletal muscle tissue biopsies will be obtained from the vastus lateralis. These samples will be analyzed by GC-MS and NMR spectroscopy to quantify the isotopomer intermediates of the TCA cycle and measure the corresponding TCA cycle flux. The flux estimations from the arteriovenous blood samples will be compared to that obtained directly from the skeletal muscle tissue. This methodology will be validated in the setting of low insulin levels alone or in combination with high glucagon concentrations.

SECONDARY OUTCOMES:
Changes in the protein and metabolite contents within circulating exosomes derived from the arterial-venous blood supply of the skeletal muscle and splanchnic tissue | 12 hours
Changes in the metabolome derived from the arterial-venous blood supply of the skeletal muscle and splanchnic tissue | 12 hours
Changes in the proteome derived from the arterial-venous blood supply of the skeletal muscle and splanchnic tissue in response to hormonal manipulation. | 12 hours
Oxygen consumption in skeletal muscle and splanchnic tissue in response to hormonal manipulation | 12 hours
Mitochondrial respiration in skeletal muscle tissue | 12 hours
Reactive oxygen species emissions in skeletal muscle tissue | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: K Sreekumaran Nair, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akram M. Citric acid cycle and role of its intermediates in metabolism. Cell Biochem Biophys. 2014 Apr;68(3):475-8. doi: 10.1007/s12013-013-9750-1. PMID 24068518
- [Background] Befroy DE, Perry RJ, Jain N, Dufour S, Cline GW, Trimmer JK, Brosnan J, Rothman DL, Petersen KF, Shulman GI. Direct assessment of hepatic mitochondrial oxidative and anaplerotic fluxes in humans using dynamic 13C magnetic resonance spectroscopy. Nat Med. 2014 Jan;20(1):98-102. doi: 10.1038/nm.3415. Epub 2013 Dec 8. PMID 24317120
- [Background] Sunny NE, Parks EJ, Browning JD, Burgess SC. Excessive hepatic mitochondrial TCA cycle and gluconeogenesis in humans with nonalcoholic fatty liver disease. Cell Metab. 2011 Dec 7;14(6):804-10. doi: 10.1016/j.cmet.2011.11.004. PMID 22152305
- [Background] Schumann WC, Magnusson I, Chandramouli V, Kumaran K, Wahren J, Landau BR. Metabolism of [2-14C]acetate and its use in assessing hepatic Krebs cycle activity and gluconeogenesis. J Biol Chem. 1991 Apr 15;266(11):6985-90. PMID 2016310
- [Background] Alves TC, Pongratz RL, Zhao X, Yarborough O, Sereda S, Shirihai O, Cline GW, Mason G, Kibbey RG. Integrated, Step-Wise, Mass-Isotopomeric Flux Analysis of the TCA Cycle. Cell Metab. 2015 Nov 3;22(5):936-47. doi: 10.1016/j.cmet.2015.08.021. Epub 2015 Sep 24. PMID 26411341
- [Background] Jones JG, Solomon MA, Cole SM, Sherry AD, Malloy CR. An integrated (2)H and (13)C NMR study of gluconeogenesis and TCA cycle flux in humans. Am J Physiol Endocrinol Metab. 2001 Oct;281(4):E848-56. doi: 10.1152/ajpendo.2001.281.4.E848. PMID 11551863
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials